CLINICAL TRIAL: NCT01271439
Title: A Phase II Study of Neoadjuvant Chemotherapy + IMRT Combined With Cetuximab in Advanced T Stage of Nasopharyngeal Carcinoma
Brief Title: Study of Chemoradiotherapy Combined With Cetuximab in Nasopharyngeal Carcinoma
Acronym: REPLACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Wenzhou Medical University (Other); The First Affiliate Hospital of Guangxi Medical College (Unknown); Xijing Hospital (Other); Hunan Cancer Hospital (Other); Jiangxi Provincial Cancer Hospital (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan University (Other); Hubei Cancer Hospital (Other); Tongji University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other); Shenzhen People's Hospital (Other); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Zhao Chong, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REPLACE
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2011-11

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cetuximab (Experimental)
  Interventions: Drug: Cetuximab

INTERVENTIONS:
Drug: Cetuximab — 400mg/m2 intravenous infusion the week before radiotherapy, 250mg/m2 intravenous infusion weekly for 6 weeks during radiotherapy
  Other Names: C225

SUMMARY:
This is an open, multicenter phase Ⅱ clinical trial. The purpose of this study is to evaluate acute toxicity and efficacy of cetuximab (C225) combined with IMRT + neoadjuvant chemotherapy in advanced T stage of nasopharyngeal carcinoma. Besides, to figure out the relationship between patient outcome and EGFR gene copy number, expression and mutation.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of nasopharyngeal carcinoma
* Range from 18～69 years old
* T3-4，N0-2，M0 (AJCC 2009)
* KPS ≥ 80
* Nonmetastatic diseases
* WBC count ≥ 4×109/L，Hemoglobin ≥ 100g/L， platelet count ≥ 100×109/L
* ALT or AST < 1.5×ULN、bilirubin < 1.5×ULN
* 0Serum creatinine < 1.5×ULN

Exclusion Criteria:

* Distance metastases
* Previously treated (surgery，chemotherapy, radiation therapy，EGFR targeted therapy or immunotherapy)
* Second malignancy within 5 years
* Precious therapy with an investigational agent
* Uncontrolled seizure disorder or other serious neurologic disease
* ≥ Grade Ш allergic reaction to any drug including in this study
* Clinically significant cardiac or respiratory disease
* Creatinine clearance < 30ml/min
* Drug or alcohol addition
* Do not have full capacity for civil acts
* Severe complication, active infection
* Concurrent immunotherapy or hormone therapy for other diseases
* Pregnancy or lactation

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2012-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
3 Month Complete Response Rate + Partial Response Rate | 3 Months
  According to RECIST (Response Evaluation Criteria in Solid Tumors) criteria, Complete response was defined as disappearance of all target lesions, Partial response was defined as at least a 30% reduction in the sum of the longest diameter of target lesions.

SECONDARY OUTCOMES:
One-year locoregional control rate | 1 year
  locoregional control rate: from the time when finish treatment to persistence or recurrence in the nasopharyngeal and/or cervical region.
Three-year locoregional control rate | 3 years
  locoregional control rate: from the time when finish treatment to persistence or recurrence in the nasopharyngeal and/or cervical region.
One-year disease free survival rate | 1 year
  disease free survival rate: from the time when finish treatment to first failure at any site.
Three-year disease free survival rate | 3 years
  disease free survival rate: from the time when finish treatment to first failure at any site.
One-year overall survival rate | 1 year
  overall survival rate: from the time when finish treatment to death of any cause.
Three-year overall survival rate | 3 years
  overall survival rate: from the time when finish treatment to death of any cause.
The relationship between 3 years overall survival rate and expression of EGFR | 3 years
  all patients must have sufficient pretreatment tumor biopsy specimens.
Use EORTC QLQ-C30(version 3.0) and EORTC QLQ-H&N35(Version 1.0) to access the quality of life | 3 years
  collect date before treatment, the week using neoadjuvant chemotherapy, every week during radiotherapy, 6 months and every year after all treatment finished.
The relationship between 3 years overall survival rate and amplification of EGFR | 3 years
  all patients must have sufficient pretreatment tumor biopsy specimens.
The relationship between 3 years overall survival rate and mutation of EGFR | 3 years
  all patients must have sufficient pretreatment tumor biopsy specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Chong Zhao, Principal Investigator — Sun Yat-sen University; Yunfeng Zhou, Principal Investigator — Zhongnan Hospital
Locations (1):
- Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Home Page of Cancer Center, Sun Yat-sen University — http://www.sysucc.org.cn